CLINICAL TRIAL: NCT06610448
Title: Wearable Evaluation of Ambulatory Readings for Blood Pressure
Acronym: WEAR-BP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stephen Juraschek (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Stephen Juraschek, Principal Investigator, Beth Israel Deaconess Medical Center
Organization: Beth Israel Deaconess Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2024P000441; 5R01HL158622 (NIH)
Record Dates: First submitted 2024-09-12; First posted 2024-09-24 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Normal Blood Pressure; Controlled Hypertension; Uncontrolled Hypertension
Keywords: Cuff-based BP device; Cuffless BP device; ABPM; Blood Pressure; Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Each participant is randomly assigned a different blood pressure device each day over the course of 3 days. All participants will use each device, but the devices will be applied on different days and on different arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (3):
- Cuff-based ambulatory blood pressure monitor sequence (Experimental): Participants will be randomized 1:1 to wear (A) the Spacelabs ambulatory blood pressure monitor on the first day and ABPMPro ambulatory blood pressure monitor on the second day or (B) ABPMPro ambulatory blood pressure monitor on the first day then Spacelabs ambulatory blood pressure monitor on the second day.
  Interventions: Device: ABPMPro; Device: Spacelabs Ambulatory Blood Pressure Monitoring
- Left versus right upper limb (Experimental): Participants will be randomized to wear the Aktiia cuffless blood pressure device on either the left upper limb versus the right upper limb on the first day. On the second day, the Aktiia blood pressure device will be switched to the other arm which did not get randomized on the first day. Another wristband (LiveMetric versus Bpro) will be worn on the contralateral arm.
  Interventions: Device: Aktiia Blood Pressure; Device: LiveMetric; Device: Bpro
- Wristband sequence (first day versus second day) (Experimental): Participants will be randomized 1:1 to wear (A) the LiveMetric wristband on the first day and Bpro wristband on the second day or (B) Bpro wristband on the first day then LiveMetric wristband on the second day. The arm side (i.e., right or left) will be determined by the Aktiia cuffless blood pressure device randomization on the first day. For the second day, the Aktiia cuffless blood pressure device will be worn on the arm opposite the first day with the other device (LiveMetric versus Bpro) worn on the contralateral arm.
  Interventions: Device: Aktiia Blood Pressure; Device: LiveMetric; Device: Bpro

INTERVENTIONS:
Device: ABPMPro — This is an upper arm, cuff-based intermittent ambulatory BP device. This device has an internal activity and body position sensor which gathers information about sleep-wake estimation.
  Arms: Cuff-based ambulatory blood pressure monitor sequence
Device: Spacelabs Ambulatory Blood Pressure Monitoring — This is an upper arm cuff-based device with tubing for continuous ambulatory BP monitoring with a unique activity sensor that correlate with patient movement activity with blood pressure changes.
  Arms: Cuff-based ambulatory blood pressure monitor sequence
Device: Aktiia Blood Pressure — This is a wrist cuff-based device which uses an optical sensor (photoplethysmography sensor) to gather data from the arteries under the skin surface. Aktiia has an upper arm cuff device which is used for calibration once every month to provide a baseline blood pressure reading.
  Arms: Left versus right upper limb; Wristband sequence (first day versus second day)
Device: LiveMetric — This is a wrist cuff-based applanation tonometry continuous ambulatory BP device. This device has automatic self-calibration and comes in various sizes.
  Arms: Left versus right upper limb; Wristband sequence (first day versus second day)
Device: Bpro — This is a wrist cuff-based wireless oscillometric, continuous ambulatory BP device. It has applanation tonometry at the wrist with Pulse wave analysis. This device needs calibration with a brachial cuff BP measurement.
  Arms: Left versus right upper limb; Wristband sequence (first day versus second day)

SUMMARY:
The purpose of this project is to compare the performance and validity of novel wearable technologies that measure blood pressure (BP) and physical activity with a Spacelabs Ambulatory Blood Pressure Monitoring (ABPM) device.

DETAILED DESCRIPTION:
The investigators will recruit community-dwelling participants to wear novel cuffless BP monitoring devices for comparison with a Spacelabs ABPM device throughout a 24-hour period. The identification of accurate cuffless BP technologies would greatly improve access to ABPM and allow for BP measurements at times when the use of cuff-based devices are not feasible. Knowledge from this project will inform subsequent research protocols among adults and under-represented groups.

Up to 250 participants (at least 100) will be involved in this study each wearing up to 7 devices (6 BP devices and 1 activity monitor). The assignment of devices will be randomized by day and by the arm or wrist on which they are worn. During the first visit, participants will provide their consent and be randomly fitted with 3 BP devices; either the Spacelabs ABPM device or the ABPMpro device, the Aktiia wristband BP monitor, and one of two other cuff-based wrist BP monitors, along with an activity monitor to track body positions. These devices will be worn continuously for at least 24-hours, including overnight, before being returned. On the following day, for Visit 2, participants will be fitted with a different set of 3 BP devices; the ABPMpro device or Spacelabs ABPM device, the Aktiia wristband BP device (on the opposite wrist from the previous day), and the final cuff-based wristband BP device. Additionally, participants will wear an ambulatory BP device as a patch on the chest. These devices will also be worn for at least 24 hours. This study will enable characterization of the feasibility, practicality, and effectiveness of the measurements and the devices' accuracy and precision.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 100 years
* All neighborhoods in Boston area
* Be able to walk with two limbs and have two arms
* Willing and able to complete required measurement procedures
* Able to provide informed consent

Exclusion Criteria:

* Failure to receive informed consent
* Arm circumference of more than 50cm

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06-06 (Actual); Primary Completion 2026-05-03 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Systolic Blood Pressure | 24 - 48 hours
  Measured from all 5 randomized devices

SECONDARY OUTCOMES:
Diastolic Blood Pressure | 24 - 48 hours
  Measured from all 5 randomized devices
Heart Rate | 24 - 48 hours
  Measured from all 5 randomized devices
ActivPaL device (Physical activity monitor) | 24 - 48 hours
  Physical activity intensity and type of activity will be characterized throughout the 48hr wear period. While the investigators are interested in the impact of devices on activity, the investigators are also interested in the relationship between activities and blood pressure.

OTHER OUTCOMES:
Systolic blood pressure from the Biobeat device (Chest Patch Blood Pressure device) | 24 hours
  This is a continuous ambulatory BP device which is worn as a patch on the chest. This device needs calibration with a brachial cuff BP measurement. This will be typically worn on day 2. This is not a randomized assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
Participants will be consented in the event data will be shared with other investigators.

REFERENCES:
- See also: Study website for potential participants — http://wearbp.org